CLINICAL TRIAL: NCT05466136
Title: Effects of Mental Fatigue on Inhibitory Control and Endurance Performance in Athletes With Different Levels of Dispositional Mindfulness: An Event-Related Potential Study
Brief Title: Mindfulness, Mental Fatigue, Inhibitory Control and Endurance Performance in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: PACNL_JT_MF_Trait
Record Dates: First submitted 2022-07-06; First posted 2022-07-20 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Mental Fatigue
Keywords: Mindfulness; Athletes; Mental fatigue; Inhibitory control; Endurance performance
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Intervention Model Description: The participants will visit the lab on two counterbalanced order occasions to complete either an incongruent version Stroop task (mental fatigue condition, MF) or a congruent version Stroop task (control condition, CON) for 30 minutes to induce the mental fatigue state.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental fatigue condition (Experimental): Performing a completed incongruent version of Stroop task for 30min.
  Interventions: Behavioral: Mental fatigue condition
- Control condition (Experimental): Performing a completed congruent version of Stroop task for 30min.
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: Mental fatigue condition — In mental fatigue condition, the mental fatigue manipulation will use a modified Stroop task with complete incongruent trials, which is wildly used to induce a mentally fatigued state in previous studies. The Stroop task included four colored words presented in traditional Chinese (i.e., red, green, blue, and yellow), the color of the word will paint inconsistent with the semantic meaning of the word (e.g., red word printed in green). The task consisted of five 6-minute blocks and 1080 incongruent trials for each block. The total duration will be 30-min.
  Arms: Mental fatigue condition
Behavioral: Control condition — Similar to mental fatigue conditions, the modified Stroop task with complete congruent trials will be used, The Stroop task also included four colored words presented in traditional Chinese (i.e., red, green, blue, and yellow), but the color of the word will paint consistent with the semantic meaning of the word (e.g., red word printed in red) in order to set up the match condition of relative less cognitive demanding for participants. Same with the mental fatigue condition, the task consisted of five 6-minute blocks and 1080 congruent trials for each block. The total duration will be 30-min.
  Arms: Control condition

SUMMARY:
This study investigated the mediating effect of dispositional mindfulness on the impact of mental fatigue on neurocognitive functions and endurance performance in athletes.

DETAILED DESCRIPTION:
Recent research suggests that mental fatigue by prolonged cognitive tasks would impair neurocognitive functions (e.g., executive functions, brain activity) and sports performance, especially inhibitory control and endurance performance. On the other hand, individuals with higher dispositional mindfulness have been linked to greater athletic performance and cognitive functions. Still, there is little known whether higher dispositional mindfulness counteracts the detrimental effects of mental fatigue on endurance performance and inhibitory control in athletes. Therefore, this study is conducted to investigate whether dispositional mindfulness mediates the effects of mental fatigue on neurocognitive functions and endurance performance in athletes.

The qualified participants will visit the lab on two counterbalanced order occasions to complete either a modified incongruent Stroop task (mental fatigue condition, MF) or a modified congruent Stroop task (control condition, CON) for 30 minutes. Before and after each cognitive task, participants will be measured for their subjective mental fatigue by a visual analog scale (VAS). After each cognitive task, inhibitory control and endurance performance will be evaluated by a Flanker task and a graded exercise test (GXT), respectively. Furthermore, the general and athletic dispositional mindfulness will be measured using the Five Facet Mindfulness Questionnaire (FFMQ) and Athlete Mindfulness Questionnaire (AMQ), respectively.

Specifically, the targeted primary outcomes are neurocognitive functions (i.e., reaction time, accuracy and ERPs in Flanker task) and endurance performance (i.e., VO2max & time to exhaustion in GXT); The secondary outcomes are subjective (i.e., VAS score)/objective (i.e., reaction time, accuracy in Stroop task) mental fatigue, motivation in tasks, mood (i.e., BRUMS-C).

ELIGIBILITY:
Inclusion Criteria:

1. Regular sports training at least 4 hours weekly
2. Normal or corrected-to-normal vision
3. Right-handed

Exclusion Criteria:

1. Physical limitation or injury in lower limbs before and during the study
2. Diagnosed or self-reported neurological disorders (e.g., epilepsy)
3. Diagnosed or self-reported major psychiatric illness (e.g., major depression, schizophrenia)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Inhibitory control: Reaction time | about 1 year
  Inhibitory control will be evaluated by a Flanker task in terms of reaction time in this study, and the types of trials are the congruent (i.e., > > > > >) and incongruent (i.e., < < > < <). In the Flanker task, participants will be presented with five arrows and will be instructed to respond as quickly and accurately as possible to the direction where the middle arrow is pointing (i.e., left or right).
Inhibitory control: Accuracy | about 1 year
  Inhibitory control will be evaluated by a Flanker task in terms of accuracy in this study, and the types of trials are the congruent (i.e., > > > > >) and incongruent (i.e., < < > < <). In the Flanker task, participants will be presented with five arrows and will be instructed to respond as quickly and accurately as possible to the direction where the middle arrow is pointing (i.e., left or right).
Endurance performance: Time to exhaustion | about 1 year
  The endurance performance in terms of time to exhaustion (TTE) will be assessed by graded exercise test (GXT) with Bruce protocol on treadmill (h/p/cosmos pulsar 3p, Germany). The initial speed and grade of the GXT will be set at 2.74 km/hr with grade of 10% and increase speed and grade every 3 min until participants are volitionally exhausted.
Endurance performance: Maximum Oxygen Consumption | about 1 year
  The maximal oxygen consumption (VO2max) throughout the whole GXT will be recorded by a computerized indirect calorimetry system (SensorMedics Vmax 29C, USA), and until the participants reached volitional exhaustion. The VO2max in the study will be defined as the highest 30-s average value of VO2 measured during GXT.
Changes in neuroelectrical activities | about 1 year
  The neuroelectrical activities during the computerized cognitive tasks (i.e., Stroop task & Flanker task) will be recorded. The changes in the event-related potential (e.g., P3) will be analyzed.

SECONDARY OUTCOMES:
Subjective mental fatigue | about 1 year
  Before, after Stroop task, and after Flanker task, changes in subjective mental fatigue will be measured using a visual analog scale for mental fatigue (VAS-MF). Participants will be asked the following questions "What is your mental fatigue level now?", and participants could indicate how mental fatigue on a scale from 0 (i.e., no mental fatigue at all) to 100 (i.e., completely mentally exhausted).
Objective mental fatigue: Reaction time in Stroop task | about 1 year
  During the intervention, the reaction time in both Stroop tasks will be calculated as an index of objective mental fatigue.
Objective mental fatigue: Accuracy in Stroop task | about 1 year
  During the intervention, the accuracy in both Stroop tasks will be calculated as an index of objective mental fatigue.
Rating of perceived exertion | about 1 year
  The Rating of perceived exertion (RPE) will be measured at beginning and every 2.5-min during the GXT using Borg 6 to 20 scale, until the participant comes to voluntary exhaustion.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, Ph.D, Study Director — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (1):
- Department of Physical Education and Sport Sciences, National Taiwan Normal University, Taipei, Taiwan